CLINICAL TRIAL: NCT01537237
Title: Randomized Comparison of Rotational Angiography/Electroanatomical Mapping Fusion Versus CT/Electroanatomical Mapping Fusion to Guide AF Ablation
Brief Title: Comparison of Rotational Angiography/Electroanatomical Mapping Fusion Versus CT/Electroanatomical Mapping Fusion to Guide AF Ablation
Acronym: 3DATGvsCT
Status: Completed | Type: Observational
Sponsor: Steward St. Elizabeth's Medical Center of Boston, Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: 00591
Record Dates: First submitted 2012-01-03; First posted 2012-02-23 (Estimated); Last update posted 2014-11-25 (Estimated); Status verified 2012-03

CONDITIONS: Atrial Fibrillation; Arrhythmia
Keywords: Atrial Fibrillation; Catheter-based ablation; Pulmonary vein isolation; Electro-anatomical mapping; Rotational angiography
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- intra-procedure 3DATG: Patients who will undergo intra-procedure 3DATG rotational angiography to guide their ablation procedure
- pre-procedure CT: Patients who will undergo pre-procedure CT scan to guide their ablation procedure

SUMMARY:
The purpose of this study is to compare rotational angiography (3DATG technology)intra-procedure (during the ablation procedure) with CT (x-ray) pre-procedure (before the ablation procedure) fusion to create an anatomical picture of a heart to help adequately guide an ablation procedure for patients with arrhythmias.

DETAILED DESCRIPTION:
Rotational angiography (or three dimensional arteriography or "3DATG") is a new tool used to guide atrial fibrillation (AF) ablation. The current approach to imaging for AF ablation involves obtaining a computer tomography (CT) angiogram of the atrium pre-procedure and combining it with an electro-anatomical map, a process called merging or overlay. The investigators propose to investigate the quality of the 3DATG as a replacement for the CT in obtaining a left atrial angiogram (to guide AF ablation).

All imaging modalities to be evaluated in this study are currently used in clinical practice. They are not experimental methods. The goal is to compare two modalities that have never been directly compared before. The CT angiography utilizes a standard CT scanner and intravenously injected contrast agent to visualize the left atrium. While the 3DATG is a method that achieves similar results to a CT scanner, the difference is that the 3DATG images are acquired by rotating the X-ray source around the patient on a C-arm instead of a dedicated CT scanner.

60 participants will be consented and randomized to either pre-procedure CT or intra-procedure 3DATG. Scheduled participants will undergo sedation and catheter instrumentation as appropriate. CT anatomy data will then be merged with the live X-ray via the EP Navigator system in standard fashion or the patient will be prepped for appropriate 3DATG anatomy data acquisition and merged with the EP Navigator system. The EP Navigator system will then be used to send either data to NavX or CARTO to create the intended electro-anatomical map.

Using the CT or 3DATG acquired electro-anatomical map, the ablation procedure will be conducted in the same way as would the local practice and standard of care for any patient not participating in the study.

The ablation procedure and the sites of ablation lesions will be tagged on the 3D overlaid anatomy in the same fashion as previously published and all participants will be followed as routine at a 1 month and 3 month follow up.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing a clinically indicated left-sided ablation procedure for atrial fibrillation

Exclusion Criteria:

* Patients not willing or able to provide consent to participate or already involved in another clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients undergoing a clinically indicated left-sided ablation procedure for atrial fibrillation who therefore satisfy conventional criteria for catheter ablation.
Sampling Method: Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2011-08; Primary Completion 2013-08 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Evidence of procedural success for an ablation procedure using 3DATG fusion | within 6 months
  Case report forms were created to capture intraprocedure data (i.e.noticeable map drift) of the maps created and used to create ablation lesions. Procedure user's overall clinical evaluation (i.e.feedback) and experience (i.e. radiation time, number of mapping points collected per map, mapping time) will also be collected and analyzed. And patients will be followed as routine for overall disease evaluation (i.e. ECG and patient reported symptoms) within 6 months from the procedure.

SECONDARY OUTCOMES:
Overall radiation exposure to the patient | Pre-procedure (for CT cohort) to end of procedure
  Case report forms were created to capture the exposure each cohort of patients will be subjected to.

CONTACTS AND LOCATIONS:
Overall Officials: Michael V Orlov, MD, PhD, Principal Investigator — St. Elizabeth's Medical Center
Locations (2):
- United States (2):
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - St. Elizabeth's Medical Center, Brighton, Massachusetts